CLINICAL TRIAL: NCT06580847
Title: Speech-in-noise, Psychosocial, and Heart Rate Variability Outcomes of Group Singing or Audiobook Club Interventions for Older Adults With Unaddressed Hearing Loss: a SingWell Project Multisite, Randomized Controlled Trial.
Brief Title: Benefits of Choir for Older Adults With Unaddressed Hearing Loss (WP2)
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Toronto Metropolitan University (Other)
Collaborators: Memorial University of Newfoundland (Other); University of Groningen (Other); Flinders University (Other); Concordia University, Montreal (Other); University of Southern California (Other); University of Oldenburg (Other); University of Nottingham (Other); The Bionics Institute of Australia (Other)
Responsible Party: Principal Investigator, Frank Russo, Principal Investigator, Toronto Metropolitan University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Multisite HL 2024-103
Record Dates: First submitted 2024-08-22; First posted 2024-08-30 (Actual); Last update posted 2025-09-18 (Actual); Status verified 2025-09

CONDITIONS: Hearing Loss, Age-Related; Speech Intelligibility; Psychosocial Functioning
Keywords: Hearing loss; speech in noise; psychosocial wellbeing
MeSH Terms: conditions — Presbycusis; Speech Intelligibility; Hearing Loss

STUDY DESIGN:
Intervention Model Description: 12 week RCT exploring the benefits of group singing and an audiobook club (1.5 hours per week)
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group Singing (Experimental): 12 week group singing program consisting of 1.5 hours of in-person choir instruction per week.
  Interventions: Behavioral: Audiobook Club
- Audiobook Club (Active Comparator): 12 week group program consisting of 1.5 hours of in-person audiobook club discussion per week.
  Interventions: Behavioral: Group Singing

INTERVENTIONS:
Behavioral: Group Singing — 12 week choir program consisting of 1.5 hours of in-person instruction per week.
  Arms: Audiobook Club
Behavioral: Audiobook Club — 12 week audiobook club program consisting of 1.5 hours of in-person discussion per week.
  Arms: Group Singing

SUMMARY:
Unaddressed age-related hearing loss is highly prevalent among older adults, typified by negative consequences for speech-in-noise perception and psychosocial wellbeing. There is promising evidence that group singing may enhance speech-in-noise perception and psychosocial wellbeing. However, there is a lack of robust evidence, primarily due to the literature being based on small sample sizes, single site studies, and a lack of randomized controlled trials. Hence, to address these concerns, this SingWell Project study utilizes an appropriate sample size, multisite, randomized controlled trial approach, with a robust preplanned statistical analysis.

The objective of the study is to explore if group singing may improve speech-in-noise perception and psychosocial wellbeing for older adults with unaddressed hearing loss.

The investigators designed an international, multisite, randomized controlled trial to explore the benefits of group singing for adults aged 60 years and older with unaddressed hearing loss. After undergoing an eligibility screening process and completing an information and consent form, the investigators intend to recruit 210 participants that will be randomly assigned to either group singing or an audiobook club (control group) intervention for a training period of 12-weeks. The study has multiple timepoints for testing, that are broadly categorized as macro (i.e., pre- and post-measures across the 12-weeks), or micro timepoints (i.e., pre- and post-measures across a weekly training session). Macro measures include behavioural measures of speech and music perception, and psychosocial questionnaires. Micro measures include psychosocial questionnaires and heart-rate variability.

The investigators hypothesize that group singing may be effective at improving speech perception and psychosocial outcomes for older adults with unaddressed hearing loss-more so than participants in the control group.

ELIGIBILITY:
Inclusion Criteria:

1. Adults aged 60 years and older;
2. Bilateral mild-to-moderate hearing loss (20-49 dB hearing level), measured using four-frequency pure-tone average across both ears (4FPTA) measured at 500 Hz, 1000 Hz, 2000 Hz, and 4000 Hz;
3. Unaddressed hearing loss (i.e., participants must not currently use a hearing aid, cochlear implant, or assistive listening device);
4. No significant cognitive impairment, to be assessed with the Montreal Cognitive Assessment for people with hearing impairment (MoCA-H), with participants requiring a score ≥ 24;
5. Not use a pacemaker or anti-arrhythmic agents/medications;
6. Not currently participating in regular active music learning (e.g., choir, formal music training) or audiobook clubs within the last year; and
7. Sufficient language capacity to understand and complete the test materials. Note: all materials will be presented written and/or aurally in English at the sites located in Canada, United States of America, and Australia; Dutch at the Netherlands site; and German at the Germany site.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 210 (Estimated)
Dates: Start 2025-04-15 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Speech-in-noise perception | Baseline and completion (week 0 and week 13)
  The Coordinate Response Matrix (CRM) generates signal-to-noise ratio (SNR). A lower SNR is indicative of better speech-in-noise perception.
Emotional speech perception | Baseline and completion (week 0 and week 13)
  The EmoHI is calculated as the mean accuracy of correct responses as a percentage (0 to 100%).
Quality of Life/Wellness | Baseline and completion (week 0 and week 13)
  The 12-item short-form survey version 2 (SF-12v2) from the Medical Outcomes Study (MOS) generates a Physical Summary and a Mental Summary of patient quality of life. Scores range from 0 to 100, where a zero score indicates the lowest level of health and 100 indicates the highest level of health.
Anxiety and Depression | Baseline and completion (week 0 and week 13)
  The Hospital Anxiety and Depression Scale (HADS) provides a score between 0 and 21, with higher scores indicative of higher levels of anxiety or depression.
Self Esteem | Baseline and completion (week 0 and week 13)
  The Collective Self-Esteem Scale (CSES) consists of four scales: Membership self-esteem, Private collective self-esteem, Public collective self-esteem, and Importance to Identity. Each scale is scored between 1 and 7, with a higher score indicating high levels of self-esteem.
Social Connectedness | Baseline and completion (week 0 and week 13)
  The revised Social Connectedness Scale (SCS-R) is scored as a total between 8 and 48 points, with higher scores indicating higher levels of social connectedness.
Pitch perception | Baseline and completion (week 0 and week 13)
  The Frequency Difference Limen (FDL) task evaluates pitch perception threshold. A lower threshold indicates better pitch perception abilities.
Rhythm perception | Baseline and completion (week 0 and week 13)
  The Beat Alignment Test (BAT) measures rhythm perception accuracy between 0 and 100%.
Timbre perception | Baseline and completion (week 0 and week 13)
  The Spectral-temporally Modulated Ripple Test (SMRT) is a proxy measure of timbre perception. It generates a threshold based on performance. A higher ripple-per-octave threshold is indicative of better spectro-temporal (timbre) perception.
Higher-level Music perception | Baseline and completion (week 0 and week 13)
  The Music-in-Noise Task (MINT) is an auditory stream segregation task that is a proxy measure of higher-level music perception. It is scored as proportion correct between 0 and 1.
Positive and Negative Affect | Pre- and post-session (week 2, 7, 11)
  The Positive and Negative Affect Schedule (PANAS) consists of a positive and negative outcome measure; each ranging between 10 and 50. For the positive scale, a higher score represents higher levels of positive affect. One the negative scale, a lower score represents lower levels of negative affect.
Anxiety and Discomfort | Pre- and post-session (week 2, 7, 11)
  The Subjective Units of Discomfort Scale (SUDS) is scored between 0 and 100, with descriptive anchor points. 0 = "no anxiety, calm, relaxed"; 25 = "mild anxiety, alert, able to cope"; 50 = "moderate anxiety, some trouble concentrating"; 75 = "severe anxiety, thoughts of leaving"; and 100 = "very severe anxiety, worst ever experienced".
Social closeness | Pre- and post-session (week 2, 7, 11)
  The Inclusion of Other in the Self Scale (IOS) is scored between 1 and 7, with a higher score representing more social closeness.

OTHER OUTCOMES:
Heart rate variability and social bonding | Pre- and post-session (week 2, 7, 11)
  Heart rate variability (HRV) is a proxy measure of social bonding. Higher HRV is anticipated to be associated with higher levels of social bonding.

CONTACTS AND LOCATIONS:
Overall Officials: Frank Russo, PhD, Study Director — Toronto Metropolitan University
Locations (7):
- Brain and Creativity Institute, University of Southern California, Los Angeles, California, United States
- Flinders University, Adelaide, South Australia, Australia
- Canada (3):
  - Memorial University of Newfoundland, St. John's, Newfoundland and Labrador
  - Toronto Metropolitan University, Toronto, Ontario
  - Concordia University, Montreal, Quebec
- Carl von Ossietzky Universitat Oldenburg, Oldenburg, Germany
- University of Groningen, Groningen, Netherlands

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lo CY, Zendel BR, Baskent D, Boyle C, Coffey E, Gagne N, Habibi A, Harding E, Keijzer M, Kreutz G, Maat B, Schurig E, Sharma M, Dang C, Gilmore S, Henshaw H, McKay CM, Good A, Russo FA. Speech-in-noise, psychosocial, and heart rate variability outcomes of group singing or audiobook club interventions for older adults with unaddressed hearing loss: A SingWell Project multisite, randomized controlled trial, registered report protocol. PLoS One. 2024 Dec 4;19(12):e0314473. doi: 10.1371/journal.pone.0314473. eCollection 2024. PMID 39630812